CLINICAL TRIAL: NCT03524079
Title: Morphological and Functional Characteristics of the Right Ventricle in Patients With Brugada Syndrome
Brief Title: Right Ventricle Morphology and Hemodynamics in BrS
Acronym: RV-BrS
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Head of Arrhythmology Department, IRCCS Policlinico S. Donato
Other Study IDs: RV & BrS
Record Dates: First submitted 2018-04-19; First posted 2018-05-14 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Lorajmine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BrS Group: Ajmaline 17-(Chloroacetate) Monohydrochloride
  Interventions: Drug: Ajmaline 17-(Chloroacetate) Monohydrochloride
- No BrS group: Ajmaline 17-(Chloroacetate) Monohydrochloride
  Interventions: Drug: Ajmaline 17-(Chloroacetate) Monohydrochloride

INTERVENTIONS:
Drug: Ajmaline 17-(Chloroacetate) Monohydrochloride — Ajmaline 17-(Chloroacetate) Monohydrochloride(1mg/kg in 5 minutes)

SUMMARY:
The study purpose is to evaluate the morphological, functional and electrophysiological characteristics of the right ventricle before and after ajmaline in patients diagnosed with Brugada syndrome as well as to correlate CMR findings and substrate size.

DETAILED DESCRIPTION:
All consecutive patients with either spontaneous or ajmaline-induced BrS-ECG pattern will be screened. A total of 30 BrS patients and 30 normal age, sex and BSA matched normal controls will be selected and enrolled. Patients will perform cardiac magnetic resonance imaging to evaluate and compare morphological and functional characteristics of the 2 groups before and after ajmaline. BrS patients will also perform a standardized programmed ventricular stimulation protocol and electroanatomical mapping to determine the substrate size.

ELIGIBILITY:
Inclusion Criteria:

* Brugada syndrome with either spontaneous or ajmaline- induced type 1 ECG pattern
* Indication to ajmaline testing and programmed ventricular stimulation
* Age > or equal to 18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Contraindication to CMRI or to ajmaline
* Live espectance < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 60 selected subjects (30 BrS patients and 30 normal controls) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Electrocardiographic changes | 1 day during Electrocardiography
  Changes of PR, QRS, and QT parameters, before and after ajmaline in Brugada patients as compared with control subjects
MRI changes of left and right ventricular function | 1day during MRI
  MRI changes of left and right ventricular function before and after ajmaline in Brugada patients as compared with control subjects
CMR parameters changes of the right and left ventricle function | 1 day during CMR
  Changes of right ventricular areal strain before and after ajmaline in Brugada patients as compared with controls
Electrical substrate changes of the right ventricle | 1 day after ICD implantation
  electroanatomical epicardial mapping for substrate determination before and after ajmaline

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — IRCCS San Donato University Hospital Policlinico San Donato, Milan, Italy
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pappone C, Santinelli V, Mecarocci V, Tondi L, Ciconte G, Manguso F, Sturla F, Vicedomini G, Micaglio E, Anastasia L, Pica S, Camporeale A, Lombardi M. Brugada Syndrome: New Insights From Cardiac Magnetic Resonance and Electroanatomical Imaging. Circ Arrhythm Electrophysiol. 2021 Nov;14(11):e010004. doi: 10.1161/CIRCEP.121.010004. Epub 2021 Oct 25. PMID 34693720